CLINICAL TRIAL: NCT04081558
Title: Follow-up of Cancer Patients Receiving Chemotherapy or Targeted Therapy by Electronic Patient Reported Outcomes-tool
Brief Title: Electronic Symptom Follow-up of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Koivunen, adjuvant professor, medical oncologist, Oulu University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OuluUH2
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic follow-up (Experimental)
  Interventions: Device: Electronic patient reported outcomes tool

INTERVENTIONS:
Device: Electronic patient reported outcomes tool — Electronic patient reported outcomes

SUMMARY:
Use of ePROs in oncological care have resulted in improvement of QoL, decreased ER visits, and improvement of overall survival. Furthermore, ePRO follow-up resulted in better QoL, improved ECOG status and more active cancer treatments at disease relapse, and improved survival among cancer survivals. The current study investigates electronic patient reported outcome tool in the follow-up of cancer patients receiving chemotherapies or targeted therapies.

The aims of the current study are: 1) The number of alerts triggered by Kaiku Cancer medical treatment side-effects questionnaire and their correlation to treatment side-effects, other relevant medical events, tumor progression, and survival 2) Changes in Kaiku QLQ-C30 QoL questionnaire and their correlation to cancer treatment response, side-effects, other relevant medical event or survival 3) Patient compliance to Kaiku ePRO surveillance during treatment period according to response rates of Patient experience survey, Kaiku Cancer medical treatment side-effects questionnaire and Kaiku QLQ-C30 QoL questionnaire

In addition, in the CRC (colorectal cancer) cohort:

1. Integration of laboratory values to patient reported symptoms when prescribing a new chemotherapy cycle
2. Number of phone calls related to prescribing a new chemotherapy cycle
3. Unscheduled doctor appointments in oncology unit
4. ER visits
5. Days in hospitalization
6. Unscheduled investigations in health care
7. Development of peripheral neurotoxicity
8. The number of chemotherapy dose reductions
9. The number of chemotherapy delays
10. Health care user experience survey

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study procedure
2. Advanced breast, lung, colorectal, or pancreatic cancer
3. New cancer medical treatment, chemotherapy or targeted therapy initiated within -/+ 2 weeks from signed consent
4. Age ≥18y
5. ECOG 0-2
6. CRC cohort: Patients with adjuvant treatment, or first or second line of treatment for metastatic disease
7. Patient compliant with study procedures

Exclusion Criteria:

1. Initiation of new cancer medical treatment > 2 wks from signed consent
2. Any medical condition that the Investigator considers significant to compromise the safety of the patient or that impairs the interpretation of study assessments
3. No internet access/email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the spectrum of patient reported symptoms | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Percentages of patient reported symptoms using KaikuHealth 15 symptom e-questionnaire. Individual questions evaluate the presence of a specific symptom e.g. nausea. Questions are answered yes or no.
Change in Patient reported symptom severity | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Percentages of patient reported symptoms and their severity according NCI-CTCAE by KaikuHealth algorithm
Change in the number of triggered alerts by the tool | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Number of triggered alerts by the tool and their correlation to treatment side-effects, cancer progression, other medical events in percentages or survival.
Changes in Quality of Life according to QLQ-C30 Summary scores | At baseline, and at 4, 8, and 12weeks
  The correlation of the Summary score of QLQ-C30 to treatment side-effects, cancer progression, or other medical events or survival.
  The Core Quality of life questionnaire (QLQ-C30) is a validated cancer health-related quality-of-life questionnaire that includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality of life and financial impact. Subjects respond on a four-point-scale from "not at all" to "very much" for most items. Raw scores are linearly converted to a 0-100 scale. For the functioning scales and global QoL higher scores indicate better functioning; for the symptom scales higher scores indicate higher symptom burden. The summary score of QLQ-C30 is calculated from the mean of 13 of 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included).
Correlation between changes in different symptoms and their severity to treatment side-effects, cancer progression, other medical events, or survival | At 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation between different patient reported symptoms and their severity to treatment side-effects, cancer progression or other medical events in percentages or survival
Changes in Patient compliance Questionnaire | At 4, 8, and 12weeks
  Patient compliance using KaikuHealth e-questionnaire addressing usability (easiness to use from scale: very easy to very difficult; need of assistance to use the program: yes/no; how understandable are questions in symptom questionnaire from scale: totally agree to totally disagree) and user experience (use of the ePRO tool will better your cancer care: yes-no, do not know; use of the ePRO tool has been useful: yes-no-do not know; would you recommend the ePRO tool for cancer care: yes-no-do not know). Analysis is done on percentages of each answer choice at specific time point(s).
Changes in patient compliance according to answering rate to symptom questionnaires | At 4, 8, and 12weeks
  Patient compliance using response rates (within one week) to symptom questionnaires in percentages from sent requests
Change in patient compliance according to answering rates to QLQ-C30 questionnaire | At 4, 8, and 12weeks
  Patient compliance using response rates to QLQ-C30 questionnaires (within one week) in percentages from sent requests. The QLQ-C30 questionnaire includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality of life and financial impact. Subjects respond on a four-point-scale from "not at all" to "very much" for most items. Raw scores are linearly converted to a 0-100 scale. For the functioning scales and global QoL higher scores indicate better functioning; for the symptom scales higher scores indicate higher symptom burden. The summary score of QLQ-C30 is calculated from the mean of 13 of 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included).

OTHER OUTCOMES:
Integration of laboratory values to patient reported symptoms when prescribing a new chemotherapy cycle in the CRC cohort | At 2-3 weeks cycle upon chemotherapy dosing schema during the treatment phase of the trial
  An integrated electronic follow-up tool combining patient reported outcomes and the results of the safety laboratory values taken before treatment
Number of phone calls related to prescribing a new chemotherapy cycle in the CRC cohort | At 2-3 weeks cycle upon chemotherapy dosing schema during the treatment phase of the trial
  Number of un-scheduled phone calls to patients from health care professionals before a new chemotherapy cycle
Unscheduled doctor appointments in oncology unit in the CRC cohort | During the treatment phase of the trial or up tp 24 weeks
  The number of unscheduled doctor appointments in oncology unit due to patient-related issues
Emergency Clinic visits in the CRC cohort | During the treatment phase of the trial or up to 24 weeks
  The number of Emergency Clinic visits
Days in hospitalization in the CRC cohort | During the treatment phase of the trial or up to 24 weeks
  The number of days in hospitalization
Unscheduled investigations in health care in the CRC cohort | During the treatment phase of the trial or up to 24 weeks
  The number of unscheduled investigations in health care
Development of peripheral neurotoxicity in the CRC cohort | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12 weeks
  The severity of peripheral neurotoxicity according to NCI-CTCAE By KaikuHealth algorithm
The number of chemotherapy dose reductions | During the treatment phase of the trial or up to 24 weeks
  The number of chemotherapy dose reductions due to patient-related issues
The number of chemotherapy delays | During the treatment phase of the trial or up to 24 weeks
  The number of chemotherapy delays due to patient-related issues
Health care user experience survey | Monthly during the treatment phase of the trial or up to 24 weeks
  A questionnaire assessing the feasibility of electronic follow-up from health care professionals point of view

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Oulu University Hospital, Oulu
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04081558/Prot_SAP_000.pdf